CLINICAL TRIAL: NCT01303861
Title: Concurrent Bupropion / Varenicline for Smoking Cessation
Acronym: ConNic4
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); Philip Morris USA, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Pro00027351; 1P50DA027840-01A1 (NIH)
Record Dates: First submitted 2011-02-23; First posted 2011-02-25 (Estimated); Results first posted 2014-08-01 (Estimated); Last update posted 2014-08-06 (Estimated); Status verified 2014-05

CONDITIONS: Nicotine Dependence
Keywords: Nicotine addiction; Cigarette smoking; Smoking cessation; Zyban; Chantix; Nicotine patches; Nicotrol Inhaler; varenicline; bupropion
MeSH Terms: conditions — Tobacco Use Disorder; Cigarette Smoking; Smoking Cessation | interventions — Varenicline; Bupropion; Tobacco Use Cessation Devices; Nicotine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- varenicline (Active Comparator): This group will consist of smokers who, based on smoking behavior, DO NOT respond favorably to pre-cessation nicotine patches (assessed at Session P2). They will receive varenicline.
  Interventions: Drug: Varenicline
- Nicotine Patches only (Active Comparator): This group will consist of smokers who, based on smoking behavior, respond favorably to pre-cessation nicotine patches(assessed at Session P2). They will continue to receive only nicotine patches.
  Interventions: Drug: Nicotine patches
- Nicotine Patches with Nicotine Inhaler (Active Comparator): This group will consist of smokers who, based on smoking behavior, respond favorably to pre-cessation nicotine patches (assessed at Session P2). They will continue to receive nicotine patches and will receive a nicotine inhaler to use as needed after their quit date.
  Interventions: Drug: Nicotine patches; Drug: Nicotine Inhaler
- varenicline with bupropion (Active Comparator): This group will consist of smokers who, based on smoking behavior, DO NOT respond favorably to pre-cessation nicotine patches (assessed at Session P2). They will receive varenicline in combination with bupropion.
  Interventions: Drug: Varenicline; Drug: Bupropion

INTERVENTIONS:
Drug: Varenicline — For the first 3 days after being switched from nicotine patches (occurring at one week before the target quit date), smokers in this group will receive varenicline at a dose of 0.5 mg once per day followed by 0.5 mg twice a day for the remaining 4 days of that week. Subsequently, the dose will be 1 mg twice per day, and will remain at that dose for the remainder of the 12 weeks.
  Other Names: Chantix
  Arms: varenicline; varenicline with bupropion
Drug: Bupropion — For the first 3 days after being switched from nicotine patches (occurring at one week before the target quit date), smokers in this group will receive bupropion at a dose of 150mg once per day. Subsequently, the dose will be 150mg twice per day, and will remain at that dose for the remainder of the 12 weeks.
  Other Names: Zyban
  Arms: varenicline with bupropion
Drug: Nicotine patches — Nicotine Replacement Therapy Groups:
  1. For smokers with high baseline carbon monoxide (CO): 42 mg/24 h for 2 weeks before the quit date and 3 weeks after the quit date, 21 mg/24 h for 4 weeks, 14 mg/24 h for 2 weeks, and 7 mg/24 h for 2 weeks; or
  2. For smokers with low baseline CO: 21 mg/24 h for 2 weeks before the quit date and 7 weeks after the quit date, 14 mg/24 h for 2 weeks, and 7 mg/ 24 h for 2 weeks.
  Varenicline and varenicline in combination with bupropion groups:
  1. For smokers with high baseline CO: 42 mg/24 h for 1 week
  2. For smokers with low baseline CO: 21 mg/24 h for 1 week
  Other Names: Nicoderm
  Arms: Nicotine Patches only; Nicotine Patches with Nicotine Inhaler
Drug: Nicotine Inhaler — Nicotine inhaler to use as needed after quit date
  Other Names: Nicotrol Inhaler
  Arms: Nicotine Patches with Nicotine Inhaler

SUMMARY:
This study focuses on the first step in developing an algorithm for maximizing quit-smoking success based on an adaptive approach, which changes treatment from the initial nicotine replacement therapy (NRT) when that treatment alone may not be sufficient. These NRT "non-responders" are switched (in double-blind fashion) before the quit date to receive either varenicline alone or varenicline paired with bupropion. Some participants who would otherwise have failed at their quit smoking attempt could be "rescued" by switching to alternative pharmacotherapies. The proposed study will evaluate the combination treatment against varenicline alone in an adaptive trial design

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years old;
* smoked an average of at least 10 cigarettes per day for three cumulative years;
* have an expired air CO reading assessed at screening of at least 10ppm;
* express a desire to quit smoking within the next 30 days.

Exclusion Criteria:

* Hypertension (systolic >140 mm Hg, diastolic >100 mm Hg, coupled with a history of hypertension); subjects with no previous diagnosis of hypertension may have a screening blood pressure up to 160/100.
* Hypotension with symptoms (systolic <90 mm Hg, diastolic <60 mm Hg).
* Coronary heart disease;
* Lifetime history of heart attack;
* Cardiac rhythm disorder (irregular heart rhythm);
* Chest pains (unless history, exam, and ECG clearly indicate a non-cardiac source);
* Cardiac (heart) disorder (including but not limited to valvular heart disease, heart murmur, heart failure);
* History of skin allergy;
* Active skin disorder (e.g., psoriasis) within the last five years, except minor skin conditions (including but not limited to facial acne, minor localized infections, and superficial minor wounds);
* Liver or kidney disorder (except kidney stones, gallstones);
* Gastrointestinal problems or disease other than gastroesophageal reflux or heartburn;
* Active ulcers in the past 30 days;
* Currently symptomatic lung disorder/disease (including but not limited to chronic obstructive pulmonary disease (COPD), emphysema, and asthma);
* Brain abnormality (including but not limited to stroke, brain tumor, and seizure disorder);
* Migraine headaches that occur more frequently than once per week;
* Recent, unexplained fainting spells;
* Problems giving blood samples;
* Diabetes treated with insulin; non-insulin treated diabetes (unless glucose is less than 180mg/dcl and HbA1c is less than 7%);
* Current cancer or treatment for cancer in the past six months (except basal or squamous cell skin cancer);
* Other major medical condition;
* Current psychiatric disease (with the exception of anxiety disorders, obsessive compulsive disorder (OCD) and ADHD);
* Suicidal ideation (within the past 10 years) or lifetime occurrence of attempted suicide;
* Current depression;
* Bulimia or anorexia;
* Pregnant or nursing mothers;
* Alcohol abuse;
* Use of Opiate medications for pain or sleep in the past 14 days;
* Significant adverse reaction to nicotine patches, nicotine inhalers, bupropion / Wellbutrin / Zyban or Chantix / Varenicline in the past.
* Use (within the past 30 days) of:
* Illegal drugs (or if the urine drug screen is positive),
* Experimental (investigational) drugs;
* Psychiatric medications including antidepressants, anti-psychotics or any other medications that are known to affect smoking cessation (e.g. clonidine);
* Smokeless tobacco (chewing tobacco, snuff), cigars, pipes or e-cigarettes;
* Wellbutrin, bupropion, Zyban, Chantix, nicotine replacement therapy or any other smoking cessation aid.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 702 (Actual)
Dates: Start 2011-03; Primary Completion 2013-03 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jed E Rose, Ph.D., Principal Investigator — Duke University
Locations (4):
- United States (4):
  - Duke Center for Nicotine and Smoking Cessation Research, Charlotte, North Carolina
  - Duke Center for Nicotine and Smoking Cessation Research, Durham, North Carolina
  - Duke Center for Nicotine and Smoking Cessation Research, Raleigh, North Carolina
  - Duke Center for Nicotine and Smoking Cessation Research, Winston-Salem, North Carolina

REFERENCES:
- [Derived] Livingstone-Banks J, Fanshawe TR, Thomas KH, Theodoulou A, Hajizadeh A, Hartman L, Lindson N. Nicotine receptor partial agonists for smoking cessation. Cochrane Database Syst Rev. 2023 May 5;5(5):CD006103. doi: 10.1002/14651858.CD006103.pub8. PMID 37142273
- [Derived] Hartmann-Boyce J, Theodoulou A, Farley A, Hajek P, Lycett D, Jones LL, Kudlek L, Heath L, Hajizadeh A, Schenkels M, Aveyard P. Interventions for preventing weight gain after smoking cessation. Cochrane Database Syst Rev. 2021 Oct 6;10(10):CD006219. doi: 10.1002/14651858.CD006219.pub4. PMID 34611902
- [Derived] Rose JE, Behm FM. Combination treatment with varenicline and bupropion in an adaptive smoking cessation paradigm. Am J Psychiatry. 2014 Nov 1;171(11):1199-205. doi: 10.1176/appi.ajp.2014.13050595. PMID 24934962

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment began on 3/07/11 and ended on 11/30/12. Of the 702 subjects consented during this period, 218 were in our Charlotte, NC office, 157 were in our Durham, NC office, 151 were in our Raleigh, NC office and 176 were in our Winston-Salem, NC office. Only 349 subjects met all study criteria, and 22 discontinued prior to being assigned.
Groups:
- Nicotine Patches Only: This group will consist of smokers who, based on smoking behavior, respond favorably to pre-cessation nicotine patches(assessed at Session P2). They will continue to receive only nicotine patches.
  Nicotine patches: Nicotine Replacement Therapy Groups:
  1. For smokers with high baseline CO: 42 mg/24 h for 2 weeks before the quit date and 3 weeks after the quit date, 21 mg/24 h for 4 weeks, 14 mg/24 h for 2 weeks, and 7 mg/24 h for 2 weeks; or
  2. For smokers with low baseline CO: 21 mg/24 h for 2 weeks before the quit date and 7 weeks after the quit date, 14 mg/24 h for 2 weeks, and 7 mg/ 24 h for 2 weeks.
  Varenicline and varenicline in combination with bupropion groups:
  1. For smokers with high baseline CO: 42 mg/24 h for 1 week
  2. For smokers with low baseline CO: 21 mg/24 h for 1 week
- Nicotine Patches With Nicotine Inhaler: This group will consist of smokers who, based on smoking behavior, respond favorably to pre-cessation nicotine patches (assessed at Session P2). They will continue to receive nicotine patches and will receive a nicotine inhaler to use as needed after their quit date.
  Nicotine patches: Nicotine Replacement Therapy Groups:
  1. For smokers with high baseline CO: 42 mg/24 h for 2 weeks before the quit date and 3 weeks after the quit date, 21 mg/24 h for 4 weeks, 14 mg/24 h for 2 weeks, and 7 mg/24 h for 2 weeks; or
  2. For smokers with low baseline CO: 21 mg/24 h for 2 weeks before the quit date and 7 weeks after the quit date, 14 mg/24 h for 2 weeks, and 7 mg/ 24 h for 2 weeks.
  Varenicline and varenicline in combination with bupropion groups:
  1. For smokers with high baseline CO: 42 mg/24 h for 1 week
  2. For smokers with low baseline CO: 21 mg/24 h for 1 week
  Nicotine Inhaler: Nicotine inhaler to use as needed after quit date
Period: Overall Study
Arm/Group | Varenicline | Nicotine Patches Only | Nicotine Patches With Nicotine Inhaler | Varenicline With Bupropion
Started | 109 | 50 | 55 | 113
Finished Treatment Phase | 71 | 34 | 39 | 72
Completed | 51 | 25 | 19 | 54
Not Completed | 58 | 25 | 36 | 59
Not completed — Lost to Follow-up | 34 | 14 | 27 | 31
Not completed — Lack of Efficacy | 3 | 2 | 1 | 0
Not completed — Withdrawal by Subject | 16 | 8 | 8 | 23
Not completed — Adverse Event | 4 | 1 | 0 | 5
Not completed — Pregnancy | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Subjects who failed to respond to pre-cessation nicotine patch treatment were randomized to receive varenicline, or varenicline + bupropion. Subjects who showed reductions in ad lib smoking were randomly assigned to nicotine patch only or patch + nicotine inhaler. 22 Subjects discontinued study participation prior to being assigned to a condition.
Groups:
- Nicotine Patches Only: This group will consist of smokers who, based on smoking behavior, respond favorably to pre-cessation nicotine patches(assessed at Session P2). They will continue to receive only nicotine patches.
  Nicotine patches: Nicotine Replacement Therapy Groups:
  1. For smokers with high baseline carbon monoxide (CO): 42 mg/24 h for 2 weeks before the quit date and 3 weeks after the quit date, 21 mg/24 h for 4 weeks, 14 mg/24 h for 2 weeks, and 7 mg/24 h for 2 weeks; or
  2. For smokers with low baseline CO: 21 mg/24 h for 2 weeks before the quit date and 7 weeks after the quit date, 14 mg/24 h for 2 weeks, and 7 mg/ 24 h for 2 weeks.
  Varenicline and varenicline in combination with bupropion groups:
  1. For smokers with high baseline CO: 42 mg/24 h for 1 week
  2. For smokers with low baseline CO: 21 mg/24 h for 1 week
- Dropped Prior to Condition Assignment: These subjects discontinued study participation prior to being assigned to a condition.
- Total: Total of all reporting groups
Arm/Group | Varenicline | Nicotine Patches Only | Nicotine Patches With Nicotine Inhaler | Varenicline With Bupropion | Dropped Prior to Condition Assignment | Total
Number analyzed (Participants) | 109 | 50 | 55 | 113 | 22 | 349
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 109 | 49 | 54 | 113 | 22 | 347
  >=65 years | 0 | 1 | 1 | 0 | 0 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.58 (11.39) | 45.20 (10.56) | 42.09 (12.22) | 44.22 (10.47) | 44.77 (11.28) | 44.42 (11.20)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 63 | 30 | 34 | 58 | 10 | 195
  Male | 46 | 20 | 21 | 55 | 12 | 154
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 1 | 1 | 2 | 1 | 9
  Not Hispanic or Latino | 105 | 49 | 54 | 111 | 21 | 340
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 0 | 0 | 1
  Asian | 2 | 0 | 0 | 0 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 0 | 0 | 1
  Black or African American | 32 | 20 | 19 | 41 | 9 | 121
  White | 71 | 29 | 31 | 68 | 11 | 210
  More than one race | 1 | 1 | 3 | 3 | 2 | 10
  Unknown or Not Reported | 3 | 0 | 0 | 1 | 0 | 4
Region of Enrollment [Number; unit: participants]
  United States | 109 | 50 | 55 | 113 | 22 | 349

OUTCOME MEASURES:

1. Primary Outcome: Four-week Continuous Abstinence From Cigarette Smoking
Description: The primary dependent measures will be continuous four-week abstinence from weeks 8-11 post target quit date, defined as a self-report of no smoking confirmed by expired air carbon monoxide.
Time Frame: Study week 8 thru week 11
Population: 1 subject from varenicline group excluded from analysis due to pregnancy. 1 subject from Nicotine Patches only group excluded due to meeting an exclusion criteria.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Varenicline | Nicotine Patches Only | Nicotine Patches With Nicotine Inhaler | Varenicline With Bupropion
Number analyzed (Participants) | 108 | 49 | 55 | 113
percentage of participants | 25.93 [17.97 to 35.25] | 46.94 [32.53 to 61.73] | 43.64 [30.30 to 57.68] | 39.82 [30.73 to 49.46]

2. Secondary Outcome: Seven Day Point Abstinence From Cigarette Smoking
Description: Secondary outcome will include point abstinence (no smoking in the previous 7-day) at 6 months post-quit.
Time Frame: Six months post quit date
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: participants
Arm/Group | Varenicline | Nicotine Patches Only | Nicotine Patches With Nicotine Inhaler | Varenicline With Bupropion
Number analyzed (Participants) | 108 | 49 | 55 | 113
participants | 18 [11 to 27] | 12 [7 to 19] | 6 [2 to 12] | 29 [20 to 39]

3. Secondary Outcome: Continuous Cigarette Abstinence From Quit Date
Description: Secondary outcome will include continuous abstinence from quit date to end of treatment (week 11).
Time Frame: From Quit date to end of treatment (week 11)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: participants
Arm/Group | Varenicline | Nicotine Patches Only | Nicotine Patches With Nicotine Inhaler | Varenicline With Bupropion
Number analyzed (Participants) | 108 | 49 | 55 | 113
participants | 9 [4 to 16] | 13 [7 to 20] | 15 [9 to 23] | 17 [10 to 26]

ADVERSE EVENTS:
Time Frame: Subjects were receiving study drugs for 13 weeks. At each study session during this period subjects completed a questionnaire about side effects. Subjects were also told to contact us between study sessions if side effects were bothersome.
Description: Twenty-two subjects discontinued study participation prior to being assigned a condition; therefore, no side effects data were collected.
Arm/Group | Varenicline | Nicotine Patches Only | Nicotine Patches With Nicotine Inhaler | Varenicline With Bupropion | Dropped Prior to Condition Assignment
Serious Adverse Events (participants affected / at risk) | 0/109 | 1/50 | 0/55 | 0/113 | 0/22
Other Adverse Events (participants affected / at risk) | 76/109 | 33/50 | 38/55 | 80/113 | 0/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Varenicline (N=109) | Nicotine Patches Only (N=50) | Nicotine Patches With Nicotine Inhaler (N=55) | Varenicline With Bupropion (N=113) | Dropped Prior to Condition Assignment (N=22)
Tightness in Chest (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Varenicline (N=109) | Nicotine Patches Only (N=50) | Nicotine Patches With Nicotine Inhaler (N=55) | Varenicline With Bupropion (N=113) | Dropped Prior to Condition Assignment (N=22)
Headache (Nervous system disorders) | 10 (12) | 5 (5) | 5 (5) | 9 (11) | 0 (0)
Nasal / Sinus Irritation (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 4 (5) | 3 (3) | 7 (7) | 0 (0)
Change in Taste (General disorders) | 7 (11) | 11 (13) | 10 (15) | 21 (34) | 0 (0)
Mouth / Throat Irritation (General disorders) | 7 (11) | 4 (4) | 2 (3) | 3 (3) | 0 (0)
Dry Mouth (General disorders) | 7 (12) | 6 (8) | 3 (7) | 15 (24) | 0 (0)
Thirst (General disorders) | 14 (26) | 6 (13) | 7 (11) | 18 (30) | 0 (0)
Coughing (Respiratory, thoracic and mediastinal disorders) | 12 (18) | 6 (9) | 3 (3) | 6 (7) | 0 (0)
Joint / Muscle Pain (Metabolism and nutrition disorders) | 9 (13) | 6 (12) | 3 (7) | 6 (8) | 0 (0)
Jaw / Neck Pain (General disorders) | 4 (4) | 2 (3) | 3 (4) | 1 (1) | 0 (0)
Heartburn (Gastrointestinal disorders) | 6 (9) | 3 (5) | 4 (4) | 6 (10) | 0 (0)
Nausea (Gastrointestinal disorders) | 8 (10) | 5 (6) | 3 (4) | 4 (5) | 0 (0)
Constipation (Gastrointestinal disorders) | 5 (9) | 1 (1) | 2 (2) | 9 (13) | 0 (0)
Irritability (Nervous system disorders) | 13 (18) | 6 (7) | 5 (8) | 10 (15) | 0 (0)
Nightmares (Nervous system disorders) | 1 (1) | 6 (9) | 0 (0) | 3 (3) | 0 (0)
Vivid Dreams (Nervous system disorders) | 13 (20) | 20 (41) | 12 (23) | 24 (56) | 0 (0)
Insomnia (Nervous system disorders) | 10 (15) | 14 (20) | 5 (6) | 18 (25) | 0 (0)
Nightmares (Nervous system disorders) | 7 (10) | 3 (4) | 1 (1) | 11 (13) | 0 (0)
Itching at Patch Site (Skin and subcutaneous tissue disorders) | 1 (1) | 12 (19) | 8 (12) | 2 (2) | 0 (0)
Anxiety (Nervous system disorders) | 0 (0) | 1 (1) | 7 (9) | 1 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No